CLINICAL TRIAL: NCT01570569
Title: Development of High-throughput Minidose Inje Cocktail Method for Simultaneous Evaluating Five Cytochrome P450 Isoforms in Human
Brief Title: Development of Minidose Inje Cocktail Method for Simultaneous Evaluating Five Cytochrome P450 Isoforms in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-152
Record Dates: First submitted 2011-12-06; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — Omeprazole; Losartan; Dextromethorphan; Midazolam; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Omeprazole (Active Comparator)
  Interventions: Drug: Omeprazole; Drug: Cocktail
- Losartan (Active Comparator)
  Interventions: Drug: Losartan; Drug: Cocktail
- Dextromethorphan (Active Comparator)
  Interventions: Drug: Dextromethorphan; Drug: Cocktail
- Caffeine (Active Comparator)
  Interventions: Drug: Cocktail; Drug: Caffeine
- Midazolam (Active Comparator)
  Interventions: Drug: Cocktail; Drug: Midazolam

INTERVENTIONS:
Drug: Omeprazole — Thirteen healthy male subjects were given oral doses of 200 μg omeprazole, 2 mg losartan and 2 mg dextromethorphan individually and in combination of five drugs (cocktail) every other days.
  Other Names: The drug was made by Yuhan corp.; The drug was exclusively made for this study.
  Arms: Omeprazole
Drug: Losartan — Thirteen healthy male subjects were given oral doses of 200 μg omeprazole, 2 mg losartan and 2 mg dextromethorphan individually and in combination of five drugs (cocktail) every other days.
  Other Names: The drug was made by Yuhan corp.; The drug was exclusively made for this study.
  Arms: Losartan
Drug: Dextromethorphan — Thirteen healthy male subjects were given oral doses of 200 μg omeprazole, 2 mg losartan and 2 mg dextromethorphan individually and in combination of five drugs (cocktail) every other days.
  Other Names: The drug was made by Yuhan corp.; The drug was exclusively made for this study.
  Arms: Dextromethorphan
Drug: Cocktail — Group A : Thirteen healthy male subjects were given oral doses of 200 μg omeprazole, 2 mg losartan and 2 mg dextromethorphan individually and in combination of five drugs (cocktail) every other days.
  Group B : Thirteen healthy male subjects received 100 μg midazolam and 2 mg caffeine individually followed by five-drugs cocktail every two days.
  Other Names: All of the drugs were made by Yuhan corp.; All of the drugs were exclusively made for this study.
Drug: Midazolam — Thirteen healthy male subjects received 100 μg midazolam and 2 mg caffeine individually followed by five-drugs cocktail every two days.
  Other Names: The drug was made by Yuhan corp.; The drug was exclusively made for this study.
  Arms: Midazolam
Drug: Caffeine — Thirteen healthy male subjects received 100 μg midazolam and 2 mg caffeine individually followed by five-drugs cocktail every two days.
  Other Names: The drug was made by Yuhan corp.; The drug was exclusively made for this study.
  Arms: Caffeine

SUMMARY:
The investigators objectives were developing mini dose five-drug cocktail regimen to evaluate potential drug-drug interactions associated with use of a cocktail of caffeine, losartan, omeprazole, dextromethorphan, and midazolam for simultaneous assessment of CYP1A2, CYP2C9, CYP2C19, CYP2D6, and CYP3A activities.

DETAILED DESCRIPTION:
The investigators objectives were developing minidose five-drug cocktail regimen to evaluate potential drug-drug interactions associated with use of a cocktail of caffeine, losartan, omeprazole, dextromethorphan, and midazolam for simultaneous assessment of CYP1A2, CYP2C9, CYP2C19, CYP2D6, and CYP3A activities.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject whose CYP2C9, CYP2C19, CYP2D6 genotype was determined

Exclusion Criteria:

* Subject who has abnormal laboratory test results

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cmax, AUC | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD, PhD, Principal Investigator — Inje University